CLINICAL TRIAL: NCT02350361
Title: A Study of Endostar Combination With Chemotherapy and Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors in Lung Cancer Rechallenging Treatment After Resistance of EGFR-TKI and Tumor Progression
Brief Title: Endostar Combination With Chemotherapy and EGFR-TKI in Lung Cancer Rechallenging Treatment After Acquired Resistance.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Li Liang, Associate chief physician, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH-LL01
Record Dates: First submitted 2015-01-12; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Lung Cancer
Keywords: endostar; angiogenesis; EGFR-TKI; lung caner
MeSH Terms: conditions — Lung Neoplasms | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endostar Arm (Experimental): Gefitinib re-challenging, oral daily use Docetaxel 60mg/m2 and Cisplatin 70mg/m2, 21 days Recombinant human endostatin 15mg/day, day 1 - 14
  Interventions: Drug: Recombinant human endostatin
- Standard Arm (Active Comparator): Gefitinib re-challenging, oral daily use Docetaxel 60mg/m2 and Cisplatin 70mg/m2, 21 days Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant human endostatin — Recombinant human endostatin 7.5mg/m2
  Other Names: Endostar
  Arms: Endostar Arm
Drug: Placebo — Placebo
  Arms: Standard Arm

SUMMARY:
Here we are going to find a method by using available multiple drugs including angiogenesis medicine - Endostar to treat lung cancer patients who acquired resistence from EGFR-TKI but have responsed to it before.

DETAILED DESCRIPTION:
Lung cancer patients who received epidermal growth factor receptor tyrosine kinase inhibitors(EGFR-TKI) will acquiring resistance to the drug. This is a study of using Endostar, an angiogentic medicine, combination with chemotherapy and EGFR-TKI in lung cancer rechallenging treatment after resistance of EGFR-TKI and progression disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologic confirmation of NSCLC with tissue diagnosis or cytologic diagnosis, whose NSCLCs are locally advanced or metastatic Stage III-B / IV adenocarcinoma, and are inoperable and incurable with radiotherapy.
* Life expectancy of at least three (3) months after the start of administration of the investigational drug.
* Eastern Cooperative Oncology Group (ECOG) performance Score 0 to 2.
* Patients with at least one tumor lesion that can accurately be measured by CT or MRI in at least one dimension with longest diameter to be recorded as no less than double the slice thickness and >=10 mm.
* Patient received at least 6 months EGFR-TKI and show tumor progress
* Adequate hematologic hepatic and renal functions based on the normal conditions of chemotherapy
* Patient signed consent form and adherence and geographic location are liable to follow up

Exclusion Criteria:

* CNS metastasis
* Active infection
* Bleeding tendency or blood coagulation dysfunction
* History of neurological or psychiatric disorders, including epilepsy, or dementia
* Pregnancy or breast-feeding women
* Organ transplant long-term use of immunosuppressive drugs
* Arrhythmia need anti-arrhythmic treatment or other risk of heart disease
* Use other targeted drugs during the research
* Other conditions may not allowed to join in this study according to the researcher's judgment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Objective Responese Rate | in two months

SECONDARY OUTCOMES:
Progression Free Survival | up to six months
Overall Survial | follow up every two months, about two years
Number of Serious Adverse Events | within two months

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China